CLINICAL TRIAL: NCT03141034
Title: Ramucirumab Plus Irinotecan in Patients With Previously Treated Advanced Gastric or Gastro-esophageal Junction Adenocarcinoma
Brief Title: Ramucirumab Plus Irinotecan for Previously Treated Advanced Gastric or Gastro-esophageal Junction Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201704082
Record Dates: First submitted 2017-04-27; First posted 2017-05-04 (Actual); Results first posted 2024-06-11 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Gastric Adenocarcinoma; Gastro-esophageal Junction Adenocarcinoma
MeSH Terms: interventions — Irinotecan; Ramucirumab; Blood Specimen Collection; Cell-Free Nucleic Acids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Irinotecan plus ramucirumab (Experimental): -Patients will receive ramucirumab intravenously on an outpatient basis at a dose of 8 mg/kg over the course of 60 minutes on Day 1 of each 14-day cycle. They will then receive irinotecan intravenously at a dose of 180 mg/m2 over the course of 90 minutes on Day 1 of each 14-day cycle.
  Interventions: Drug: Irinotecan; Drug: Ramucirumab; Genetic: Blood for angiome profiling; Genetic: Blood for cfDNA

INTERVENTIONS:
Drug: Irinotecan — -Irinotecan is commercially available and will be billed to insurance.
  Other Names: Camptosar®; CPT-11
Drug: Ramucirumab — -Ramucirumab will be provided free of charge by Eli Lilly and Company.
  Other Names: Cyramza®
Genetic: Blood for angiome profiling — -Before treatment on cycle 1 day 1, cycle 5 day 1, cycle 9 day 1, and end of treatment
Genetic: Blood for cfDNA — -Before treatment on cycle 1 day 1, cycle 3 day 1, cycle 5 day 1, cycle 7 day 1, cycle 9 day 1, and end of treatment

SUMMARY:
The investigators hypothesize that this combination regimen of irinotecan plus ramucirumab administered as second line treatment will be tolerated and lead to improved outcomes similar to paclitaxel plus ramucirumab in patients with advanced gastric and gastro-esophageal junction (GEJ) cancers. This study proposes a phase II clinical trial with irinotecan plus ramucirumab for treatment of patients with metastatic gastric and GEJ adenocarcinoma who have progressed after first line chemotherapy. To the knowledge of the investigators, this regimen has not been previously administered to this patient population, so safety and tolerability will be monitored and reported.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically or cytologically confirmed diagnosis of gastric or gastroesophageal junction (GEJ) adenocarcinoma that is metastatic or locally advanced and unresectable.
* Measurable disease defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 10 mm with CT scan (or MRI at the discretion of the principal investigator (PI)), as ≥ 20 mm by chest x-ray, or ≥ 10 mm with calipers by clinical exam.
* Either primary or non-osseous metastatic site amenable for research biopsy for patients enrolled at Washington University, if safe and feasible, as confirmed by scheduling of biopsy procedure. Other methods to obtain appropriate cancer cells such as large-volume paracentesis or thoracentesis can be allowed at PI discretion. Biopsy or other procedures should be performed at least 7 days prior to C1D1.
* Experienced documented objective radiographic or clinical disease progression during first-line therapy or within 4 months after the last dose of first-line therapy with any platinum/fluoropyrimidine doublet with or without anthracycline (epirubicin or doxorubicin) or taxane (docetaxel) for unresectable or metastatic disease.

NOTE: This is not intended to be an exclusive list of allowed agents. The targeted therapies such as Herceptin and ADC, or immunotherapies without cytotoxic chemotherapy, are permitted.

* At least 18 years of age.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
* Normal bone marrow and organ function as defined below:

  * Absolute neutrophil count (ANC) ≥ 1,500/µL
  * Hemoglobin ≥ 9.0 g/dL (5.58 mmol/L)
  * Platelets ≥ 100,000/µL
  * Total bilirubin ≤ 1.5 mg/dL (25.65 µmol/L)
  * AST(SGOT)/ALT(SGPT) ≤ 3.0 x institutional upper limit of normal (IULN) (or ≤ 5.0 x IULN in the setting of liver metastases)
  * Creatinine ≤ 1.5 x IULN OR creatinine clearance ≥ 40 mL/min/1.73 m2 for patients with creatinine levels > 1.5 x IULN (that is, if serum creatinine is > 1.5 x IULN, a 24-hour urine collection to calculate creatinine clearance must be performed)
  * Urinary protein ≤ 1+ on dipstick or routine urinalysis (UA); if dipstick or routine UA is ≥ 2+, a 24-hour urine collection for protein must demonstrate < 1000 mg of protein in 24 hours
  * Adequate coagulation function as defined by INR ≤ 1.5 and PTT ≤ 5 seconds above the ULN (unless receiving anticoagulation therapy). Patients receiving warfarin must be switched to low molecular weight heparin and have achieved stable coagulation profile prior to first dose of protocol therapy.
  * All clinically significant toxic effects (except peripheral neuropathy) of prior locoregional therapy, surgery, or other anticancer therapy have resolved to ≤ Common Terminology Criteria for Adverse Events (CTCAE) grade 1.
  * Women of childbearing potential and men must agree to use two forms of adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately. Women of childbearing potential must have a negative serum pregnancy test within 7 days of study entry.
  * Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Squamous cell or undifferentiated gastric cancer.
* Received any chemotherapy (including irinotecan) other than platinum and fluoropyrimidine with or without anthracycline or taxane for advanced gastric or GEJ adenocarcinoma.
* Received previous systemic chemotherapy with a cumulative dose of > 900 mg/m^2 of epirubicin or > 400 mg/m^2 of doxorubicin.
* Received any previously systemic therapy (including investigational agents) targeting VEGF or the VEGFR signaling pathways. Other previous targeted therapies are permitted if stopped at least 28 days prior to start of treatment.
* A history of other malignancy ≤ 3 years previous with the exception of basal cell or squamous cell carcinoma of the skin which were treated with local resection only or carcinoma in situ of the cervix or other solid tumors treated curatively and without evidence of recurrence.
* Currently receiving any other investigational agents.
* History or evidence of known brain metastases or carcinomatous meningitis. Patients with known brain metastases must be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to monoclonal antibody treatment, any components used in the ramucirumab DP preparation, irinotecan, or other agents used in the study.
* Any grade 3-4 GI bleeding within 3 months prior to enrollment.
* History of gastrointestinal perforation and/or fistulae within 6 months prior to enrollment.
* History of deep vein thrombosis, pulmonary embolism, or any other significant thromboembolism (venous port of catheter thrombosis or superficial venous thrombosis are not considered "significant") during the 3 months prior to enrollment.
* History of any arterial thromboembolic event, including but not limited to myocardial infarction, transient ischemic attack, cerebrovascular accident, or unstable angina within 6 months prior to enrollment.
* Diagnosis of symptomatic congestive heart failure (NYHA II-IV) or symptomatic or poorly controlled cardiac arrhythmia.
* Uncontrolled or poorly controlled hypertension (> 160 mmHg systolic or > 100 mmHg diastolic for > 4 weeks) despite standard medical management.
* Presence of serious or nonhealing wound, ulcer, or bone fracture within 28 days prior to enrollment.
* Major surgery within 28 days prior to first dose of protocol therapy.
* Minor surgery/subcutaneous venous access device placement within 7 days prior to first dose of protocol therapy.
* Receiving chronic antiplatelet therapy, including aspirin, nonsteroidal anti-inflammatory drugs (NSAIDs, including ibuprofen, naproxen, and others), dipyridamole or clopidogrel, or similar agents. Once-daily aspirin use (maximum dose 325 mg/day) is permitted.
* The patient has elective or planned major surgery to be performed during the course of the clinical trial.
* Bowel obstruction, history or presence of inflammatory enteropathy or extensive intestinal resection (hemicolectomy or extensive small intestine resection with chronic diarrhea), Crohn's disease, ulcerative colitis, or chronic diarrhea.
* Cirrhosis at a level of Child-Pugh B (or worse) or cirrhosis (any degree) and a history of hepatic encephalopathy or clinically meaningful ascites resulting from cirrhosis (i.e. ascites from cirrhosis requiring diuretics or paracentesis). Patients with ascites not related to cirrhosis, such as malignant ascites, are allowed.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, metabolic disorders or other nonmalignant organ or systemic disease or secondary effects of cancer that induce a high medical risk and make assessment of survival uncertain, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and/or breastfeeding.
* Known HIV-positivity on combination antiretroviral therapy because of the potential for pharmacokinetic interactions with ramucirumab and irinotecan. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2023-04-14 (Actual); Study Completion 2023-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kian-Huat Lim, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (4):
- United States (4):
  - University of Miami - Sylvester Comprehensive Cancer Center, Miami, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Inc., Tampa, Florida
  - Washington University School of Medicine, St Louis, Missouri
  - UT Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Irinotecan Plus Ramucirumab
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Irinotecan Plus Ramucirumab
Number analyzed (Participants) | 40
Age, Continuous [Median (Full Range); unit: years] | 63 [27 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 36
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 33
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: -PFS will be measured from date of study entry to first radiographic progression or death due to any cause. Radiographic progressive disease (PD) will be defined using Response Evaluation Criteria in Solid Tumors v1.1 (RECIST v1.1). For those who are alive and do not experience progression, the investigators will censor them at the time of loss to follow-up or at 30 months from the study entry, whichever comes first.
Time Frame: Up to 30 months from completion of treatment (up to 36 months)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Irinotecan Plus Ramucirumab
Number analyzed (Participants) | 40
months | 5.257 [2.957 to 6.341]

2. Secondary Outcome: Overall Survival (OS)
Description: -OS time will be measured from date of study entry to date of death from any cause. For those who are alive, the investigators will censor them at the time of loss to follow-up or at 30 months from the date of treatment discontinuation, whichever comes first.
Time Frame: Up to 30 months from completion of treatment (estimated to be 36 months)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Irinotecan Plus Ramucirumab
Number analyzed (Participants) | 40
months | 8.51 [6.8010 to 12.518]

3. Secondary Outcome: Time to Progressive Disease (TTP)
Description: -TTP is defined as the time from study entry until date of radiographic PD using RECIST v1.1 criteria. For those who are alive and do not experience progression, the investigators will censor them at the time of loss to follow-up or at 30 months from the study entry, whichever comes first. For those who are dead before progression, the investigators will consider death as the competing risk. If the number of death are very small, the investigators will censor them at time of death.
Time Frame: Up to 30 months from completion of treatment (estimated to be 36 months)
Population: 2 participants were not evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Irinotecan Plus Ramucirumab
Number analyzed (Participants) | 38
months | 5.454 [2.957 to 7.261]

4. Secondary Outcome: Best Overall Response (BOR)
Description: -BOR is defined as the best response across all time points from randomization until radiologically confirmed PD using RECIST, v1.1 criteria. Complete response defined as the disappearance of all target and non-target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm and normalization of tumor marker level of non-target lesions. Partial response defined as having a ≥30% decrease in sum of longest diameter (LD) of target lesions. Progressive disease defined as having a ≥20% increase in sum of LD of target lesions and ≥5 mm increase above nadir. Stable disease defined as small changes that did not meet above criteria.
Time Frame: Up to end of treatment (estimated to be 6 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Irinotecan Plus Ramucirumab
Number analyzed (Participants) | 40
Participants
  Complete response | 1
  Partial response | 8
  Stable disease | 17
  Progressive disease | 6
  Not evaluable | 8

5. Secondary Outcome: Objective Response Rate (ORR)
Description: -ORR defined as confirmed complete response + confirmed partial response. Complete response defined as the disappearance of all target and non-target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm and normalization of tumor marker level of non-target lesions. Partial response defined as having a ≥30% decrease in sum of longest diameter (LD) of target lesions.
Time Frame: Up to end of treatment (estimated to be 6 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Irinotecan Plus Ramucirumab
Number analyzed (Participants) | 40
Participants | 9

6. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: -CBR defined as percentage of combined participants who have achieved confirmed complete response, confirmed partial response, and stable disease. Complete response defined as the disappearance of all target and non-target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm and normalization of tumor marker level of non-target lesions. Partial response defined as having a ≥30% decrease in sum of longest diameter (LD) of target lesions. Stable disease defined as small changes that did not meet above criteria nor the criteria for progressive disease.
Time Frame: Up to end of treatment (estimated to be 6 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Irinotecan Plus Ramucirumab
Number analyzed (Participants) | 40
Participants | 26

7. Secondary Outcome: Toxicity and Tolerability of Regimen as Measured by the Count of the Worst Grade of Adverse Event Experienced by Each Participant
Description: -The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for all toxicity reporting.
Time Frame: Up to 30 days following completion of treatment (median length of follow-up 131.5 days, full range 15-687 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Irinotecan Plus Ramucirumab
Number analyzed (Participants) | 40
Participants
  Grade 1-2 anemia | 29
  Grade 3 anemia | 1
  Grade 1-2 enlarged lymph node in groin | 1
  Grade 1-2 atrial fibrillation | 1
  Grade 1-2 palpitations | 1
  Grade 1-2 RBBB gallop splits | 1
  Grade 1-2 ear pain | 1
  Grade 1-2 vertigo | 1
  Grade 1-2 blurred vision | 1
  Grade 1-2 cataract | 1
  Grade 1-2 abdominal cramping | 2
  Grade 1-2 abdominal distension | 1
  Grade 1-2 abdominal pain | 17
  Grade 1-2 anal fissure | 1
  Grade 1-2 anal fistula | 1
  Grade 1-2 ascites | 3
  Grade 1-2 bloating | 1
  Grade 1-2 colitis | 1
  Grade 1-2 constipation | 12
  Grade 1-2 diarrhea | 24
  Grade 3 diarrhea | 3
  Grade 1-2 dry mouth | 2
  Grade 1-2 dyspepsia | 6
  Grade 1-2 dysphagia | 5
  Grade 3 dysphagia | 1
  Grade 1-2 early satiety | 1
  Grade 1-2 epigastric pain | 1
  Grade 5 esophageal hemorrhage | 1
  Grade 1-2 flatulence | 1
  Grade 1-2 gastroesophageal reflux disease | 1
  Grade 1-2 gum bleeding | 1
  Grade 1-2 hemorrhoids | 2
  Grade 1-2 hypersalivation | 1
  Grade 1-2 mucositis oral | 5
  Grade 1-2 nausea | 23
  Grade 3 nausea | 2
  Grade 1-2 oral hemorrhage | 1
  Grade 1-2 oral pain | 2
  Grade 1-2 painful bowel movement | 1
  Grade 1-2 rectal hemorrhage | 2
  Grade 1-2 stomach pain | 5
  Grade 1-2 toothache | 1
  Grade 1-2 upper gastrointestinal hemorrhage | 1
  Grade 1-2 vomiting | 16
  Grade 3 vomiting | 2
  Grade 1-2 boil type lesion on left groin | 1
  Grade 1-2 chills | 7
  Grade 1-2 edema limbs | 10
  Grade 1-2 fatigue | 24
  Grade 3 fatigue | 4
  Grade 1-2 fever | 2
  Grade 1-2 flu-like symptoms | 1
  Grade 1-2 infusion related reaction | 4
  Grade 3 infusion related reaction | 1
  Grade 1-2 injection site reaction | 1
  Grade 1-2 night sweats | 1
  Grade 1-2 non-cardiac chest pain | 5
  Grade 1-2 tardive dyskinesia | 1
  Grade 3 anaphylaxis | 1
  Grade 1-2 abdominal infection | 2
  Grade 3 bacteremia | 1
  Grade 1-2 bronchial infection | 1
  Grade 1-2 G-tube infection | 1
  Grade 1-2 gum infection (bloody gums) | 1
  Grade 1-2 hand sore infection | 1
  Grade 1-2 infection, source unknown | 1
  Grade 1-2 lung infection | 1
  Grade 3 lung infection | 1
  Grade 1-2 mucosal infection | 1
  Grade 1-2 nail infection (ingrown fingernail) | 1
  Grade 1-2 nail infection | 1
  Grade 1-2 upper respiratory infection | 2
  Grade 1-2 bruising | 2
  Grade 1-2 fall | 1
  Grade 1-2 alanine aminotransferase increased | 9
  Grade 1-2 alkaline phosphatase increased | 13
  Grade 3 alkaline phosphatase increased | 1
  Grade 1-2 aspartate aminotransferase increased | 10
  Grade 1-2 blood bilirubin increased | 2
  Grade 3 blood bilirubin increased | 1
  Grade 1-2 creatinine increased | 4
  Grade 1-2 lymphocyte count decreased | 18
  Grade 3 lymphocyte count decreased | 5
  Grade 1-2 lymphocyte count increased | 1
  Grade 1-2 neutrophil count decreased | 7
  Grade 3-4 neutrophil count decreased | 8
  Grade 1-2 platelet count decreased | 16
  Grade 1-2 weight loss | 5
  Grade 3 weight loss | 2
  Grade 1-2 white blood cell decreased | 17
  Grade 3 white blood cell decreased | 6
  Grade 1-2 anorexia | 17
  Grade 3 anorexia | 1
  Grade 1-2 dehydration | 1
  Grade 1-2 hypercalcemia | 1
  Grade 1-2 hyperglycemia | 8
  Grade 1-2 hyperkalemia | 5
  Grade 1-2 hypermagnesemia | 1
  Grade 1-2 hypernatremia | 5
  Grade 1-2 hypoalbuminemia | 22
  Grade 1-2 hypocalcemia | 9
  Grade 1-2 hypoglycemia | 5
  Grade 1-2 hypokalemia | 7
  Grade 3 hypokalemia | 1
  Grade 1-2 hyponatremia | 5
  Grade 3 hyponatremia | 1
  Grade 1-2 hypophosphatemia | 1
  Grade 1-2 vitamin D deficiency | 1
  Grade 1-2 arthralgia | 3
  Grade 1-2 back pain | 5
  Grade 1-2 bone pain | 1
  Grade 1-2 exostosis | 1
  Grade 1-2 left groin pain | 1
  Grade 1-2 generalized muscle weakness | 1
  Grade 1-2 muscle weakness lower limb | 1
  Grade 1-2 myalgia | 1
  Grade 1-2 pain in extremity | 1
  Grade 3 cognitive disturbance | 1
  Grade 5 death due to disease progression | 1
  Grade 4 disease progression | 1
  Grade 1-2 dizziness | 11
  Grade 1-2 dysgeusia | 4
  Grade 1-2 headache | 14
  Grade 1-2 peripheral motor neuropathy | 1
  Grade 3 peripheral motor neuropathy | 1
  Grade 1-2 peripheral sensory neuropathy | 2
  Grade 1-2 seizure | 2
  Grade 1-2 stroke | 1
  Grade 1-2 anxiety | 3
  Grade 1-2 confusion | 1
  Grade 3 delirium | 1
  Grade 1-2 depression | 5
  Grade 1-2 insomnia | 7
  Grade 1-2 acute kidney injury | 1
  Grade 1-2 dysuria | 1
  Grade 1-2 elevated white blood cell count in urine | 1
  Grade 1-2 hematuria | 1
  Grade 3 hematuria | 1
  Grade 1-2 proteinuria | 11
  Grade 3 proteinuria | 1
  Grade 1-2 urinary incontinence | 1
  Grade 1-2 cough | 1
  Grade 1-2 dyspnea | 8
  Grade 1-2 epistaxis | 5
  Grade 1-2 hiccups | 2
  Grade 1-2 laryngeal inflammation | 1
  Grade 1-2 nasal congestion | 2
  Grade 1-2 postnasal drip | 1
  Grade 5 respiratory failure | 1
  Grade 1-2 runny nose | 1
  Grade 1-2 sinus disorder | 1
  Grade 1-2 sore throat | 4
  Grade 1-2 alopecia | 16
  Grade 1-2 dry skin | 1
  Grade 1-2 erythema | 1
  Grade 1-2 hyperhidrosis | 2
  Grade 1-2 lesion on left leg | 1
  Grade 1-2 palmar plantar erythrodysesthesia syndrome | 1
  Grade 1-2 pruritus | 2
  Grade 1-2 rash acneiform | 2
  Grade 1-2 rash maculo-papular | 2
  Grade 1-2 rash on chest | 1
  Grade 1-2 razor burn | 1
  Grade 1-2 sweating | 2
  Grade 1-2 scalp pain | 1
  Grade 1-2 flushing | 1
  Grade 1-2 hematoma | 1
  Grade 1-2 hypertension | 7
  Grade 3-4 hypertension | 7
  Grade 1-2 hypotension | 3
  Grade 1-2 thromboembolic event | 3
  Grade 3 thromboembolic event | 4

ADVERSE EVENTS:
Time Frame: All-cause mortality was collected through completion of follow-up (up to a total of 36 months). Serious adverse events and adverse events were collected from start of treatment through 30 days following the last day of study treatment (median follow-up 131.5 days, full range 15-687 days).
Arm/Group | Irinotecan Plus Ramucirumab
All-Cause Mortality (participants affected / at risk) | 37/40
Serious Adverse Events (participants affected / at risk) | 23/40
Other Adverse Events (participants affected / at risk) | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Irinotecan Plus Ramucirumab (N=40)
Atrial fibrillation (Cardiac disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Esophageal hemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Fatigue (General disorders) | 1
Infusion related reaction (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Bacteremia (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Alkaline phosphtase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Weight loss (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Death due to disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cognitive disturbance (Nervous system disorders) | 1
Confusion (Nervous system disorders) | 1
Delirium (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Hypertension (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Irinotecan Plus Ramucirumab (N=40)
Anemia (Blood and lymphatic system disorders) | 30
Enlarged lymph node groin (Blood and lymphatic system disorders) | 1
Palpitations (Cardiac disorders) | 1
RBBB gallop splits (Cardiac disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Blurred vision (Eye disorders) | 1
Cataract (Eye disorders) | 1
Abdominal cramping (Gastrointestinal disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 17
Anal fissure (Gastrointestinal disorders) | 1
Anal fistula (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 2
Bloating (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 12
Diarrhea (Gastrointestinal disorders) | 26
Dry mouth (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 6
Dysphagia (Gastrointestinal disorders) | 5
Early satiety (Gastrointestinal disorders) | 1
Epigastric pain (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Gum bleeding (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 2
Hypersalivation (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 22
Oral hemorrhage (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 2
Painful bowel movement (Gastrointestinal disorders) | 1
Rectal hemorrhage (Gastrointestinal disorders) | 2
Stomach pain (Gastrointestinal disorders) | 5
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 15
Chills (General disorders) | 7
Edema limbs (General disorders) | 10
Fatigue (General disorders) | 27
Fever (General disorders) | 2
Flu like symptoms (General disorders) | 1
Infusion related reaction (General disorders) | 4
Injection site reaction (General disorders) | 1
Night sweats (General disorders) | 1
Non-cardiac chest pain (General disorders) | 4
Tardive dyskinesis (General disorders) | 1
Anaphylaxis (Immune system disorders) | 1
Abdominal infection (Infections and infestations) | 2
Bronchial infection (Infections and infestations) | 1
Finger nail infection (ingrown) (Infections and infestations) | 1
G-tube infection (Infections and infestations) | 1
Gum infection (bloody) (Infections and infestations) | 1
Hand sore infection (Infections and infestations) | 1
Infection, source unknown (Infections and infestations) | 1
Lung infection (Infections and infestations) | 2
Muscosal infection (Infections and infestations) | 1
Nail infection (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 1
Bruising (Injury, poisoning and procedural complications) | 2
Alanine aminotransferase increased (Investigations) | 9
Alkaline phosphatase increased (Investigations) | 13
Aspartate aminotransferase increased (Investigations) | 10
Blood bilirubin increased (Investigations) | 2
Creatinine increased (Investigations) | 4
Lymphocyte count decreased (Investigations) | 23
Lymphocyte count increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 15
Platelet count decreased (Investigations) | 16
Weight loss (Investigations) | 6
White blood cell decreased (Investigations) | 23
Anorexia (Metabolism and nutrition disorders) | 17
Dehydration (Metabolism and nutrition disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 8
Hyperkalemia (Metabolism and nutrition disorders) | 5
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 22
Hypocalcemia (Metabolism and nutrition disorders) | 9
Hypoglycemia (Metabolism and nutrition disorders) | 5
Hypokalemia (Metabolism and nutrition disorders) | 8
Hyponatremia (Metabolism and nutrition disorders) | 5
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Left groin pain (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 11
Dysgeusia (Nervous system disorders) | 4
Headache (Nervous system disorders) | 14
Peripheral motor neuropathy (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 2
Seizure (Nervous system disorders) | 1
Stroke (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 3
Depression (Psychiatric disorders) | 5
Insomnia (Psychiatric disorders) | 7
Dysuria (Renal and urinary disorders) | 1
Elevated WBC count in urine (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 12
Urinary incontinence (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Runny nose (Respiratory, thoracic and mediastinal disorders) | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 16
Boil type lesion - left groin (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2
Lesion on left leg (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysesthesia (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Rash on chest (Skin and subcutaneous tissue disorders) | 1
Razor burn (Skin and subcutaneous tissue disorders) | 1
Scalp pain (Skin and subcutaneous tissue disorders) | 1
Sweating (Skin and subcutaneous tissue disorders) | 2
Flushing (Vascular disorders) | 1
Hematoma (Vascular disorders) | 1
Hypertension (Vascular disorders) | 13
Hypotension (Vascular disorders) | 3
Thromboembolic event (Vascular disorders) | 4
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-10): https://cdn.clinicaltrials.gov/large-docs/34/NCT03141034/Prot_SAP_000.pdf